CLINICAL TRIAL: NCT00994903
Title: Prospective, Double-Blinded, Multi-Centred, Randomised Controlled Trial of Perioperative Simvastatin Use in Elective Colorectal Surgery
Brief Title: Simvastatin in Colorectal Surgery
Acronym: StatCol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Counties Manukau Health (Other); Waitemata District Health Board (Other Government); Auckland District Health Board (Other Government)
Responsible Party: Principal Investigator, Andrew G Hill, Professor Andrew Hill, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: StatCol
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Intestinal Neoplasm; Perioperative Care
Keywords: Statin; Colon; Colorectal; Intestinal Neoplasms; ERAS; Perioperative Care
MeSH Terms: conditions — Intestinal Neoplasms | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablets (Inert calcium lactate)
  Interventions: Drug: Placebo
- Simvastatin (Experimental): 40mg of Simvastatin given 3-7 days pre-op and continued till 14 days post-op
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — 40mg orally, given 3-7 days pre-op and continued till 14 days post-op
  Arms: Simvastatin
Drug: Placebo — Placebo (Inert calcium lactate) tablets 3-7 days pre-op to 14 days post-op (as per experimental arm)
  Arms: Placebo

SUMMARY:
Statins (HMG-CoA reductase inhibitors) are a widely used class of cholesterol-lowering drugs that have an established role in the medical management of cardiovascular disease. Their benefits have also been shown in the surgical setting with decreased cardiovascular complications and lower perioperative mortality following cardiac and vascular surgery. There is now considerable evidence showing statins have useful pleiotropic properties that extend beyond cholesterol lowering, including anti-inflammatory, anti-oxidant, immunomodulatory and fibrinolytic effects. Growing evidence suggests these effects may be useful in attenuating the proinflammatory and metabolic stress response to surgery and the benefit of statins may extend to other surgical settings such as abdominal surgery.

Laboratory studies demonstrate the surgically-relevant benefits of statins and show they decrease peritoneal inflammation, reduce the severity of intestinal ischaemia-reperfusion injury, improve survival in models of abdominal sepsis, decrease the formation of postoperative intraperitoneal adhesions and improve the healing of colonic anastomoses. Retrospective clinical studies show statins improve outcomes in sepsis, reduce the postoperative systemic inflammatory response syndrome (SIRS) and are associated with decreased rates of surgical wound infections and postoperative respiratory complications following various non-cardiac general surgical procedures. However, no prospective studies have specifically evaluated the perioperative use of statins in abdominal surgery. Using colorectal surgery as a model for major abdominal surgery, the investigators will conduct a randomised controlled trial evaluating the effect of perioperative statin use on postoperative morbidity, local and systemic inflammatory response, and functional recovery after surgery.

ELIGIBILITY:
Inclusion criteria:

* Consecutive consenting patients undergoing elective colectomy, rectal resection, and reversal of Hartmann's procedure at Middlemore Hospital, Manukau Surgery Centre, Auckland City Hospital, and North Shore Hospital.

Exclusion criteria:

* Acute presentation
* Already taking statins or other lipid-lowering medication
* Known adverse reaction to statins
* Hepatic dysfunction
* Moderate to severe renal dysfunction
* Previous history of rhabdomyolysis
* On contraindicated medication
* Pregnancy
* Breastfeeding
* Patient choice.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Total complications | Up to post-operative day 30
  Complications pre-defined and graded by the Clavien-Dindo classification

SECONDARY OUTCOMES:
Peritoneal Cytokines | Postoperative Day 1
Serum cytokines | Post-operative Day 1
Change in serum C-reactive protein (CRP) | Baseline and Postoperative Day 1, 2 and 3
Change in functional recovery | Baseline and Postoperative Day 1, 3, 7, 14, and 30

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Hill, MBChB MD FRACS, Principal Investigator — University of Auckland, New Zealand
Locations (3):
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Manukau Surgical Centre, Middlemore Hospital, Auckland
  - North Shore Hospital, Auckland

REFERENCES:
- [Derived] Singh PP, Lemanu DP, Soop M, Bissett IP, Harrison J, Hill AG. Perioperative Simvastatin Therapy in Major Colorectal Surgery: A Prospective, Double-Blind Randomized Controlled Trial. J Am Coll Surg. 2016 Aug;223(2):308-320.e1. doi: 10.1016/j.jamcollsurg.2016.04.004. Epub 2016 Apr 13. PMID 27086089